CLINICAL TRIAL: NCT02404675
Title: High Dose Icotinib in Advanced Non-small Cell Lung Cancer With EGFR 21 Exon Mutation (INCREASE): a Randomized, Open-label Study
Brief Title: High Dose Icotinib in Advanced Non-small Cell Lung Cancer With EGFR 21 Exon Mutation
Acronym: INCREASE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKTN-NSCLC-01
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: NSCLC
MeSH Terms: interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 21 icotinib (250mg) (Experimental): Patients with EGFR 21 exon positive are randomly assigned to higher dose icotinib group to receive icotinib with a dose of 250 mg three times per day, till progressive disease or unaccepted toxicity.
  Interventions: Drug: icotinib
- 21 icotinib (125mg) (Active Comparator): Patients with EGFR 21 exon positive are randomly assigned to routine dose icotinib group to receive icotinib with a dose of 125 mg three times per day, till progressive disease or unaccepted toxicity
  Interventions: Drug: icotinib
- 19 icotinib (125mg) (Experimental): Patients with EGFR del 19 exon positive are assigned to routine dose icotinib group to receive icotinib with a dose of 125 mg three times per day, till progressive disease or unaccepted toxicity
  Interventions: Drug: icotinib

INTERVENTIONS:
Drug: icotinib
  Other Names: conmana

SUMMARY:
This randomized, open-label study is aimed to evaluate the efficacy of high-dose icotinib in treating advanced non-small cell lung cancer patients with positive EGFR 21 exon mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB/IV lung cancer(exclude patients confirmed by sputum cytology)
* Positive EGFR 21 exon mutation or 19 exon deletion
* Age 18-75 years old with performance status of 0 to 2
* With a measurable disease(longest diameters >=10mm with Spiral computed tomography (CT)and >=20mm with conventional CT) according to RECIST Criteria
* Adequate hematological, biochemical and organ functions.

Exclusion Criteria:

* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.
* Evidence of interstitial lung diseases
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12 months

SECONDARY OUTCOMES:
Overall survival | 20 months
Objective response rates | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chest Hospital, Capital Medical University, Beijing, China